CLINICAL TRIAL: NCT07356804
Title: Biomarkers in Pediatric Inflammatory Rheumatic Diseases
Acronym: BIRPED
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-BIR-2017-97
Record Dates: First submitted 2018-11-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2018-11

CONDITIONS: Juvenile Idiopathic Arthritis; Flare Up, Symptom
Keywords: Calprotectin; Biomarkers
MeSH Terms: conditions — Arthritis, Juvenile; Symptom Flare Up

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Calprotectine — Determination of calprotectin and amyloid protein in the serum of patients

SUMMARY:
A prospective study is proposed to serially determine new biomarkers: Calprotectin and Serum Amyloid Protein, alongside 'conventional' biomarkers: CRP and ESR, to help evaluate their utility in routine clinical practice

DETAILED DESCRIPTION:
Pediatric inflammatory rheumatic diseases are relatively uncommon, but they represent the largest group of chronic diseases in childhood/adolescence and the leading cause of disability among children in developed countries. Poor control of the inflammatory activity of any of the aforementioned diseases can lead to growth failure (issues with growth and maturation), alterations in quality of life and school schedule for the patients, limitations secondary to joint impairments (especially in the case of JIA), and in the long term, the development of acquired amyloidosis (AA), which is a complication of any uncontrolled inflammatory process and significantly increases the morbidity and mortality of affected patients.The prognosis of pediatric inflammatory rheumatic diseases depends on the proper control of inflammation as well as the management of the immunosuppressive drugs used for this purpose. Even today, clinicians face many uncertainties in assessing the inflammatory status of our patients. Therefore, a prospective study is proposed to serially measure new biomarkers-Calprotectin and Serum Amyloid Protein-alongside 'conventional' biomarkers-CRP and ESR-to help evaluate their utility in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

Patients in follow-up in our Pediatric Rheumatology Unit, with the diagnoses of: Juvenile Idiopathic Arthritis, Connective Diseases or Autoinflammatory Diseases

Exclusion Criteria:

No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in follow-up in our Pediatric Rheumatology Unit, with the diagnoses of: Juvenile Idiopathic Arthritis, Connective Diseases or Autoinflammatory Diseases
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Serum Calprotectin in pediatric population with rheumatological inflammatory diseases | Months 3, 6, 9 and 12
  To assess the clinical usefulness ofserum Calprotectin in pediatric population with rheumatological inflammatory diseases

SECONDARY OUTCOMES:
Serum Amyloid Protein in pediatric population with rheumatological inflammatory diseases | Months 3, 6, 9 and 12
  To assess the clinical usefulness of Serum Amyloid Protein in pediatric population with rheumatological inflammatory diseasesSedimentation Rate and the Clinical Criterion.
  Describe the evolution over time of these markers.
Correlation biomarkers | 1 year
  Describe the correlation of Serum calportectin and Serum Amyloid Protein with the C-Reactive Protein, the Globular

CONTACTS AND LOCATIONS:
Overall Officials: Berta Magallares, Principal Investigator — Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau - IIB Sant Pau
Locations (1):
- Santa Creu i Sant Pau Hospital, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No